CLINICAL TRIAL: NCT05316597
Title: Do Terpenes Play a Role in the Stress-reducing Effects of a Forest Bathing Intervention?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Gregory Bratman, Assistant Professor: Environmental and Forest Sciences, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00013134; R21AT011242 (NIH)
Record Dates: First submitted 2022-03-09; First posted 2022-04-07 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Monoterpene Exposure During a Forest Bathing Intervention
MeSH Terms: interventions — Forest Therapy

STUDY DESIGN:
Intervention Model Description: Participants are assigned to both arms in random order
Who Masked: Participant, Investigator
Masking Description: Participants and research staff conducting the intervention will be masked to the exposure
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Terpenes On (Experimental): Forest bathing intervention with no filtration of terpenes from inhaled air using PAPR with particle-only filter ("terpenes on")
  Interventions: Behavioral: Forest bathing
- Terpenes Off (Active Comparator): Forest bathing intervention with filtration of terpenes from inhaled air using PAPR with activated charcoal filter ("terpenes off")
  Interventions: Behavioral: Forest bathing

INTERVENTIONS:
Behavioral: Forest bathing — Participants will be seated in a forest environment for an hour-long exposure to the forest

SUMMARY:
This pilot study evaluates the role terpenes play in the stress-reducing effects of a forest bathing intervention. Participants will participate in two interventions in random order: 1) terpene exposure and 2) no terpene exposure.

DETAILED DESCRIPTION:
The investigators will use an individual-level crossover design in which each session is conducted independently and on different days. Participants will be outfitted with a powered air purifying respirator (PAPR) to selectively modulate exposure to a natural suite of forest-derived volatile organic compounds (VOCs) while present in forest environments. Each participant will undergo two forest bathing sessions, one in which VOCs are not filtered (treatment condition), and one in which they are filtered (control condition). Sessions will be separated by a washout period of at least 8 days for each participant, and order will be counterbalanced. The investigators will estimate the average effect of treatment over 40 distinct treatment days against 40 distinct control/filtered days. The power and sample size calculations (N = 40) were determined using previous nature exposure studies of similar cross-over design. The study is adequately powered assuming the conventional targets of α = 0.05 and β = 0.80 with a 10% anticipated dropout rate, and including temperature, wind, and light variability during treatment days.

The specific aim of this project is to 1) assess whether VOC inhalation regulates increases in the high frequency (HF) (ms2) component of heart rate variability (HRV) as the primary outcome (with decreases in blood pressure, heart rate, self-reported stress, and levels of inflammatory cytokines in serum included as secondary outcomes); and 1a) assess the degree of association of absorbed dose of six forest-derived VOCs (i.e., α-pinene, β-pinene, β-myrcene, Δ-3-carene, limonene, β- carophyllene) in serum with these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Non-smoker
* Physically capable of walking for approximately 15-20 min from the study vehicle to the clinic and experimental locations.

Exclusion Criteria:

* Pregnancy
* Current or prior diagnosis of neurologic, hypertensive, psychiatric, respiratory disorder, or anosmia/hyposmia
* Some types of medication.
* Olfactory sensitivity threshold (assessed via UPSIT® test kit (Sensonics International, Haddon Heights, NJ)

At enrollment, participants will complete a baseline survey on demographics, personality traits, and regular nature contact and perceptions. Study staff will also use the clinically-validated UPSIT® test kit (Sensonics International, Haddon Heights, NJ) to evaluate olfactory sensitivity and identify/exclude participants with undiagnosed smell loss.

Study staff will work with participants to schedule their forest bathing sessions and review instructions on how to prepare (e.g., by avoiding alcohol, marijuana, and certain foods, drinks, and household cleaning products with high terpene concentrations 24 hrs before their session).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2023-09-21 (Actual); Study Completion 2023-09-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Bratman, PhD, Principal Investigator — University of Washington
Locations (1):
- Pack Forest, Eatonville, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Terpenes On, Then Terpenes Off: Participants first received a forest bathing session with no filtration of terpenes from inhaled air ("terpenes on") in a forest environment for an hour-long exposure to the forest. After a washout period of at least eight days, they then received a forest bathing session with filtration of terpenes from inhaled air ("terpenes off") in a forest environment for an hour-long exposure to the forest.
- Terpenes Off, Then Terpenes On: Participants first received a forest bathing session with filtration of terpenes from inhaled air ("terpenes off") in a forest environment for an hour-long exposure to the forest. After a washout period of at least eight days, they then received a forest bathing session of no filtration of terpenes from inhaled air ("terpenes on") in a forest environment for an hour-long exposure to the forest.
Period: First Session
Arm/Group | Terpenes On, Then Terpenes Off | Terpenes Off, Then Terpenes On
Started | 21 | 22
Completed | 21 | 21
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Washout Period
Arm/Group | Terpenes On, Then Terpenes Off | Terpenes Off, Then Terpenes On
Started | 21 | 21
Completed | 18 | 13
Not Completed | 3 | 8
Not completed — Lost to Follow-up | 1 | 2
Not completed — Physician Decision | 1 | 1
Not completed — Excluded before second session | 1 | 1
Not completed — Withdrawal by Subject | 0 | 4
Period: Second Session
Arm/Group | Terpenes On, Then Terpenes Off | Terpenes Off, Then Terpenes On
Started | 18 | 13
Completed | 18 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Terpenes On, Then Terpenes Off: Participants first received a forest bathing session with no filtration of terpenes from inhaled air ("terpenes on") in a forest environment during an hour-long exposure to the forest. After a washout period of at least eight days, they then received a forest bathing session with filtration of terpenes from inhaled air ("terpenes off") in a forest environment during an hour-long exposure to the forest.
- Terpenes Off, Then Terpenes On: Participants first received a forest bathing session with no filtration of terpenes from inhaled air ("terpenes on") in a forest environment during an hour-long exposure to the forest. After a washout period of at least eight days, they then received a forest bathing session with filtration of terpenes from inhaled air ("terpenes off") during a forest environment for an hour-long exposure to the forest.
- Total: Total of all reporting groups
Arm/Group | Terpenes On, Then Terpenes Off | Terpenes Off, Then Terpenes On | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.0 (14.2) | 37.1 (14.5) | 35.1 (14.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 7 | 10 | 17
  Female | 12 | 10 | 22
  Prefer to self-describe/non-binary | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 3 | 5
  Not Hispanic or Latino | 19 | 19 | 38
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 21 | 22 | 43

OUTCOME MEASURES:

1. Primary Outcome: Changes in the HF (ms^2) Component of HRV
Description: Assess whether VOC inhalation regulates psychophysiological outcomes of the terpenes-on vs. terpenes-off sessions.
  Ln High Frequency Heart Rate Variability at T2 (20 minutes into duration of exposure for each session)
Time Frame: At time point 2 (20 minutes into duration of exposure for Session 1 and Session 2 (which occurred at least 8 days after Session 1)).
Population: Participants who participated in at least one session were included in analyses though some participant data were missing due to temporary equipment failure (e.g., mobile physiology) or sample collection obstacles (e.g., serum).
Measure: Mean (Standard Deviation); unit: ms^2
Groups:
- Terpenes On: Participants when exposed to terpenes during their forest exposure session.
- Terpenes Off: Participants when not exposed to terpenes during their forest exposure session.
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 27 | 32
ms^2 | 6.65 (1.33) | 6.48 (1.14)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.914, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Mean Difference (Final Values) = 0.01

2. Secondary Outcome: Blood Pressure (Diastolic in mmHg)
Description: Assessed using mobile physiology equipment Diastolic blood pressure at T4 (60 minutes of exposure)
Time Frame: At time point 4 (60 minutes into duration of exposure for Session 1 and Session 2 (which occurred at least 8 days after Session 1)).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 30 | 37
mmHg | 75.4 (9.86) | 73.2 (11.1)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = .554, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Mean Difference (Final Values) = 1.13

3. Secondary Outcome: Beats Per Minute (BPM)
Description: Assessed using mobile physiology equipment BPM at time point 4 (60 minutes of exposure)
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 30 | 37
BPM | 61.4 (11.9) | 63.0 (13.7)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.905, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Mean Difference (Final Values) = 0.13

4. Secondary Outcome: Skin Conductance (μS)
Description: Assessed using mobile physiology equipment Skin conductance levels at time point 2 (20 minutes into exposure)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microsiemens (µS)
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 31 | 37
microsiemens (µS) | 3.28 (3.76) | 4.14 (5.94)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.076, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Mean Difference (Final Values) = -0.84
Statistical Analysis 2: Comparison: Terpenes On vs Terpenes Off; Exploratory ANOVA results comparing full and reduced models to test the effect of terpene exposure on pattern of outcome over time; Test type: Superiority; p = 0.02, ANOVA — Threshold of P < 0.05 for significance. ANCOVA results of comparing reduced vs. full model over time

5. Secondary Outcome: Self-reported Positive Affect
Description: Assessed using the shortened Positive and Negative Affect Schedule (PANAS) Positive affect at time point 2 (20 minutes of exposure) Higher scale scores are indicative of better outcome Range 5-50
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 32 | 36
Score on a scale | 12.1 (4.00) | 11.3 (4.38)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.210, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Mean Difference (Final Values) = 0.70
Statistical Analysis 2: Comparison: Terpenes On vs Terpenes Off; [analysis description as in outcome 4, analysis 2]; Test type: Superiority; p = 0.57, ANOVA — Threshold of P < 0.05 for significance. ANCOVA results of comparing reduced vs. full model over time

6. Secondary Outcome: Self-reported Stress
Description: Assessed using a single-item self report non-validated scale Self-reported stress at time point 2 (20 minutes of exposure) Higher scale score indicative of worse outcome Range 1-5
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 32 | 36
Score on a scale | 1.09 (0.390) | 1.17 (0.447)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.921, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Mean Difference (Final Values) = 0.01
Statistical Analysis 2: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.82, ANOVA — Threshold of P < 0.05 for significance. ANCOVA results of comparing reduced vs. full model over time

7. Secondary Outcome: Self-reported Negative Affect
Description: Assessed using the shortened Positive and Negative Affect Schedule (PANAS) Negative affect at time point 2 (20 minutes of exposure) Higher score on scale indicative of worse outcome Range 5-50
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 32 | 36
Score on a scale | 5.13 (0.421) | 5.31 (0.749)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.265, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Mean Difference (Final Values) = -0.16
Statistical Analysis 2: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.63, ANOVA — Threshold of P < 0.05 for significance. ANCOVA results of comparing reduced vs. full model over time

8. Secondary Outcome: Levels of CRP
Description: Assessed using blood serum collected via standard clinical methods. CRP levels at time point 4 (60 minutes of exposure).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 21 | 27
mg/L | 9.99 (7.83) | 13.4 (12.5)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.724, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Median Difference (Final Values) = -0.34

9. Secondary Outcome: Levels of Cortisol in Serum (ng/mL)
Description: Assessed using blood serum collected via standard clinical methods Cortisol levels at time point 4 (60 minutes of exposure).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 21 | 27
ng/mL | 98.6 (43.6) | 109.0 (60.0)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.716, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Mean Difference (Final Values) = -2.85

10. Secondary Outcome: Blood Pressure (Systolic in mmHg)
Description: Assessed using mobile physiology equipment Systolic blood pressure at T4 (60 minutes of exposure)
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 30 | 37
mmHg | 123 (16.9) | 121 (14.0)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.852, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Mean Difference (Final Values) = -0.53

11. Secondary Outcome: Level of TNF-alpha
Description: Assessed using blood serum collected via standard clinical methods TNF-alpha levels at time point 4 (60 minutes of exposure).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 21 | 27
pg/mL | 3.80 (2.71) | 4.27 (2.84)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.166, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Mean Difference (Final Values) = -0.79

12. Secondary Outcome: Levels of Il-6
Description: Assessed using blood serum collected via standard clinical methods IL-6 levels at time point 4 (60 minutes of exposure).
Time Frame: as for outcome 2
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 21 | 27
pg/mL | 0.547 (0.609) | 0.763 (0.820)
Statistical Analysis 1: Comparison: Terpenes On vs Terpenes Off; Test type: Superiority; p = 0.046, Mixed Models Analysis — a priori threshold for statistical significance = p < 0.05; Control for that session's baseline included in the mixed model; Mean Difference (Final Values) = -0.19

13. Other Pre Specified Outcome: Degree of Association of Sum Composite of Absorbed Dose of VOCs in Serum (μg/mL)
Description: Assess the association of absorbed dose (µg/mL) of forest-derived VOCs in serum with primary and secondary outcomes.
Time Frame: Time point 4 (60 min) for absorbed dose associations with same time point for DBP, SBP, Cortisol, Il-6, TNF-alpha, and CRP; and associations with Time point 2 (20 minutes) for HRV, SCL, positive affect, negative affect, self-reported stress, heart rate.
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: correlation coefficient
Groups:
- All Participants: Reported associations of absorbed dose of terpenes in serum with primary and secondary outcomes for all participants grouped together.
Arm/Group | All Participants
Number analyzed (Participants) | 38
correlation coefficient
  Ln-HR HRV | 1.06 [-0.38 to 2.5]
  SCL | -7.31 [-14.6 to -0.03]
  DBP | 11.89 [-4.65 to 28.42]
  SBP | 17.55 [-7.77 to 42.88]
  HR | 7.16 [-5.8 to 20.11]
  PA | 3.75 [-3.6 to 11.09]
  NA | 0.15 [-1.11 to 1.4]
  Self-reported stress | -0.38 [-1.66 to 0.89]
  Cortisol | -45.45 [-150.06 to 59.17]
  Il-6 | -0.60 [-1.63 to 0.43]
  TNF-alpha | -5.73 [-10.95 to -0.51]
  CRP | -0.70 [-1.64 to 0.25]

14. Primary Outcome: Baseline HF (ms^2) Component of HRV
Description: Assess whether VOC inhalation regulates psychophysiological outcomes of the terpenes-on vs. terpenes-off sessions.
  Ln High Frequency Heart Rate Variability at baseline.
Time Frame: At baseline (pre-exposure)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ms^2
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 28 | 33
ms^2 | 6.48 (1.40) | 6.34 (1.55)

15. Secondary Outcome: Baseline Blood Pressure (Diastolic in mmHg)
Description: Assessed using mobile physiology equipment Diastolic blood pressure at baseline.
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 32 | 37
mmHg | 67.8 (10.8) | 66.1 (11.0)

16. Secondary Outcome: Beats Per Minute (BPM)
Description: Assessed using mobile physiology equipment BPM at baseline.
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: BPM
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 32 | 37
BPM | 66.3 (13.0) | 66.6 (13.3)

17. Secondary Outcome: Skin Conductance (μS)
Description: Assessed using mobile physiology equipment Skin conductance levels at baseline.
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: microsiemens (µS)
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 31 | 36
microsiemens (µS) | 3.58 (3.94) | 3.84 (5.14)

18. Secondary Outcome: Self-reported Positive Affect
Description: Assessed using the shortened Positive and Negative Affect Schedule (PANAS) Positive affect at baseline Higher scale scores are indicative of better outcome Range 5-50
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 31 | 36
Score on a scale | 12.0 (3.74) | 12.2 (4.59)

19. Secondary Outcome: Self-reported Stress
Description: Assessed using a single-item self report non-validated scale Self-reported stress at baseline Higher scale score indicative of worse outcome Range 1-5
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 27 | 30
Score on a scale | 1.44 (0.698) | 1.57 (0.817)

20. Secondary Outcome: Self-reported Negative Affect
Description: Assessed using the shortened Positive and Negative Affect Schedule (PANAS) Negative affect at baseline Higher score on scale indicative of worse outcome Range 5-50
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 31 | 36
Score on a scale | 5.81 (1.11) | 5.92 (1.46)

21. Secondary Outcome: Levels of CRP
Description: Assessed using blood serum collected via standard clinical methods. CRP levels at baseline
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 23 | 28
mg/L | 9.93 (6.43) | 13.6 (13.7)

22. Secondary Outcome: Levels of Cortisol in Serum (ng/mL)
Description: Assessed using blood serum collected via standard clinical methods Cortisol levels at baseline
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 23 | 28
ng/mL | 117 (57.8) | 124 (55.1)

23. Secondary Outcome: Blood Pressure (Systolic in mmHg)
Description: Assessed using mobile physiology equipment Systolic blood pressure at baseline
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 32 | 37
mmHg | 119 (12.4) | 117 (13.9)

24. Secondary Outcome: Level of TNF-alpha
Description: Assessed using blood serum collected via standard clinical methods TNF-alpha levels at baseline
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 23 | 28
pg/mL | 4.03 (2.75) | 3.72 (2.64)

25. Secondary Outcome: Levels of Il-6
Description: Assessed using blood serum collected via standard clinical methods IL-6 levels at baseline
Time Frame: At baseline (pre-exposure).
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Terpenes On | Terpenes Off
Number analyzed (Participants) | 23 | 28
pg/mL | 0.585 (0.569) | 0.591 (0.776)

ADVERSE EVENTS:
Time Frame: Monitoring from pre-exposure time (i.e., meeting participants for each session, driving to forest location, application of physiology equipment, serum collection, and self-report assessments (total of ~2-4 hours)) through duration of 60 min forest exposure sessions and subsequent period after session completion (i.e., debriefing, and returning of participants from forest session location to initial meeting point (total of ~1.5-2.5 hours)).
Description: Definitions do not differ.
Arm/Group | Terpenes On | Terpenes Off
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/43
Other Adverse Events (participants affected / at risk) | 0/43 | 0/43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT05316597/Prot_000.pdf
  • Statistical Analysis Plan (2024-05-07): https://cdn.clinicaltrials.gov/large-docs/97/NCT05316597/SAP_001.pdf
  • Informed Consent Form (2023-07-25): https://cdn.clinicaltrials.gov/large-docs/97/NCT05316597/ICF_002.pdf